CLINICAL TRIAL: NCT02243059
Title: Contrast Enhanced Diffusion-weighted Magnetic Resonance Imaging for Detection of Pathologic Lymph Nodes in Ovarian Cancer - a Feasibility Study.
Brief Title: Magnetic Resonance Imaging for Lymph Node Staging in Ovarian Cancer
Acronym: MILO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Problems with availability of study medicine in clinical center
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 142030
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2014-09

CONDITIONS: Ovarian Neoplasms
Keywords: Magnetic Resonance Imaging; Gadofosveset trisodium; Nodal imaging
MeSH Terms: conditions — Ovarian Neoplasms | interventions — gadofosveset trisodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GDF-MRI (Experimental): In this pilot study, all included patients will undergo conventional MRI with contrast enhancement (gadofosveset trisodium) and diffusion weighted MRI.
  Ablavar™ solution contains 244 mg/mL (0.25 mmol/mL) gadofosveset trisodium. 0.03 mmol/kg of gadofosveset will be administered by manual injection as a single intravenous bolus injection over a period of time up to 30 seconds followed by a 25-30 ml saline flush. In practice, this comes down to the maximum of one vial for one patient (one vial contains 10 ml solution, which contains a total of 2.50 mmol of gadofosveset trisodium equivalent to 2.27 g of gadofosveset).
  Interventions: Drug: Gadofosveset trisodium (Ablavar™ ); Device: MRI

INTERVENTIONS:
Drug: Gadofosveset trisodium (Ablavar™ )
  Other Names: Ablavar; MS-325
Device: MRI

SUMMARY:
Advanced epithelial ovarian cancer has high morbidity and mortality. Patients presenting with advanced stage ovarian cancer often have cancer spread to regional lymph nodes. Imaging strategies to depict involved lymph nodes are currently not successful. The purpose of this study is to evaluate if magnetic resonance imaging (MRI) with gadofosveset trisodium contrast enhancement (GDF-MRI) and diffusion weighted imaging (DW-MRI) is able to identify involved lymph nodes in a preoperative setting. This could guide the surgeon during surgery to dissect lymph nodes which could lead to an optimal diagnosis/staging with the lowest possible morbidity. We want to determine the optimal imaging settings and feasibility of MRI for the detection of pathological lymph nodes in women with advanced (FIGO stage IIB-IV) ovarian cancer undergoing primary debulking surgery and compare this to conventional imaging with computer tomography (CT).

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant female
* Expected FIGO stage IIB-IV epithelial ovarian carcinoma
* Scheduled for primary debulking surgery
* Written informed consent
* At least 18 years of age.

Exclusion Criteria:

* Patients estimated to have more benefit from neoadjuvant chemotherapy
* Ineligibility to undergo MRI

  * Non-MR compatible metallic implants or foreign bodies (ferromagnetic aneurysm clip, pacemaker, neurostimulation system, etcetera).
  * Claustrophobia
* Ineligibility to receive gadofosveset contrast (history of contrast allergy,

  * History of a prior allergic reaction to the active substance or to any of the excipients of Ablavar™.
  * Impaired kidney function (Glomerular Filtration Rate <30 ml/min/1.73m2).
* Previous para-aortic or pelvic lymphadenectomy
* History of a malignant tumour.
* Pregnant or lactating patients. Incapacitated subjects

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of MRI in depicting lymph nodes. | One year
  Primary outcome measure is to determine the optimal imaging settings and feasibility of MRI combined with DW-MRI and GDF-MRI (gadofosveset-MRI) in the identification of pathologic lymph nodes in women with advanced stage epithelial ovarian cancer.

SECONDARY OUTCOMES:
Diagnostic accuracy of MRI. | One year
  Sensitivity, specificity, positive predictive value and negative predictive value for the detection of metastatic lymph nodes will be calculated for MRI (+/- DW-MRI and GDF-MRI) and compared with conventional CT imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Toon Van Gorp, Dr, Principal Investigator — University Hospital Maastricht / GROW
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Background] Pereira A, Magrina JF, Rey V, Cortes M, Magtibay PM. Pelvic and aortic lymph node metastasis in epithelial ovarian cancer. Gynecol Oncol. 2007 Jun;105(3):604-8. doi: 10.1016/j.ygyno.2007.01.028. Epub 2007 Feb 23. PMID 17321572
- [Background] Morice P, Joulie F, Camatte S, Atallah D, Rouzier R, Pautier P, Pomel C, Lhomme C, Duvillard P, Castaigne D. Lymph node involvement in epithelial ovarian cancer: analysis of 276 pelvic and paraaortic lymphadenectomies and surgical implications. J Am Coll Surg. 2003 Aug;197(2):198-205. doi: 10.1016/S1072-7515(03)00234-5. PMID 12892797
- [Background] Hoskins WJ, McGuire WP, Brady MF, Homesley HD, Creasman WT, Berman M, Ball H, Berek JS. The effect of diameter of largest residual disease on survival after primary cytoreductive surgery in patients with suboptimal residual epithelial ovarian carcinoma. Am J Obstet Gynecol. 1994 Apr;170(4):974-9; discussion 979-80. doi: 10.1016/s0002-9378(94)70090-7. PMID 8166218
- [Background] Kim HS, Ju W, Jee BC, Kim YB, Park NH, Song YS, Kim SC, Kang SB, Kim JW. Systematic lymphadenectomy for survival in epithelial ovarian cancer: a meta-analysis. Int J Gynecol Cancer. 2010 May;20(4):520-8. doi: 10.1111/IGC.0b013e3181d6de1d. PMID 20686371
- [Background] Maggioni A, Benedetti Panici P, Dell'Anna T, Landoni F, Lissoni A, Pellegrino A, Rossi RS, Chiari S, Campagnutta E, Greggi S, Angioli R, Manci N, Calcagno M, Scambia G, Fossati R, Floriani I, Torri V, Grassi R, Mangioni C. Randomised study of systematic lymphadenectomy in patients with epithelial ovarian cancer macroscopically confined to the pelvis. Br J Cancer. 2006 Sep 18;95(6):699-704. doi: 10.1038/sj.bjc.6603323. Epub 2006 Aug 29. PMID 16940979
- [Background] Onda T, Yoshikawa H, Yokota H, Yasugi T, Taketani Y. Assessment of metastases to aortic and pelvic lymph nodes in epithelial ovarian carcinoma. A proposal for essential sites for lymph node biopsy. Cancer. 1996 Aug 15;78(4):803-8. doi: 10.1002/(SICI)1097-0142(19960815)78:43.0.CO;2-Z. PMID 8756375
- [Background] Kumar Dhingra V, Kand P, Basu S. Impact of FDG-PET and -PET/CT imaging in the clinical decision-making of ovarian carcinoma: an evidence-based approach. Womens Health (Lond). 2012 Mar;8(2):191-203. doi: 10.2217/whe.11.91. PMID 22375721
- [Background] Wakefield JC, Downey K, Kyriazi S, deSouza NM. New MR techniques in gynecologic cancer. AJR Am J Roentgenol. 2013 Feb;200(2):249-60. doi: 10.2214/AJR.12.8932. PMID 23345344
- [Background] Lin G, Ho KC, Wang JJ, Ng KK, Wai YY, Chen YT, Chang CJ, Ng SH, Lai CH, Yen TC. Detection of lymph node metastasis in cervical and uterine cancers by diffusion-weighted magnetic resonance imaging at 3T. J Magn Reson Imaging. 2008 Jul;28(1):128-35. doi: 10.1002/jmri.21412. PMID 18581404
- [Background] Yamashita T, Takahara T, Kwee TC, Kawada S, Horie T, Inomoto C, Hashida K, Yamamuro H, Myojin K, Luijten PR, Imai Y. Diffusion magnetic resonance imaging with gadofosveset trisodium as a negative contrast agent for lymph node metastases assessment. Jpn J Radiol. 2011 Jan;29(1):25-32. doi: 10.1007/s11604-010-0513-2. Epub 2011 Jan 26. PMID 21264658
- [Background] Low RN, Barone RM. Combined diffusion-weighted and gadolinium-enhanced MRI can accurately predict the peritoneal cancer index preoperatively in patients being considered for cytoreductive surgical procedures. Ann Surg Oncol. 2012 May;19(5):1394-1401. doi: 10.1245/s10434-012-2236-3. PMID 22302265
- [Background] Lambregts DM, Beets GL, Maas M, Kessels AG, Bakers FC, Cappendijk VC, Engelen SM, Lahaye MJ, de Bruine AP, Lammering G, Leiner T, Verwoerd JL, Wildberger JE, Beets-Tan RG. Accuracy of gadofosveset-enhanced MRI for nodal staging and restaging in rectal cancer. Ann Surg. 2011 Mar;253(3):539-45. doi: 10.1097/SLA.0b013e31820b01f1. PMID 21239980
- [Background] Schipper RJ, Smidt ML, van Roozendaal LM, Castro CJ, de Vries B, Heuts EM, Keymeulen KB, Wildberger JE, Lobbes MB, Beets-Tan RG. Noninvasive nodal staging in patients with breast cancer using gadofosveset-enhanced magnetic resonance imaging: a feasibility study. Invest Radiol. 2013 Mar;48(3):134-9. doi: 10.1097/RLI.0b013e318277f056. PMID 23262788